CLINICAL TRIAL: NCT05886920
Title: A Phase 1/2, Open Label, Dose-escalation, and Dose-expansion Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Recommended Phase 2 Dose of D3S-002 Monotherapy or Combination Therapy in Adult Subjects With Advanced Solid Tumors With MAPK Pathway Mutations
Brief Title: A Phase 1/2 Study of D3S-002 as Monotherapy or Combination Therapy in Adult Subjects With Advanced Solid Tumors With MAPK Pathway Mutations
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: D3 Bio (Wuxi) Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D3S-002-100
Record Dates: First submitted 2023-05-24; First posted 2023-06-02 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumors With MAPK Pathway Mutations
Keywords: Advanced solid tumors; mitogen-activated protein kinase; mutation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- D3S-002 Monotherapy (Experimental): Part 1: Dose Escalation, D3S-002 administered orally.
  Interventions: Drug: D3S-002
- D3S-002 and D3S-001 Combination Therapy (Experimental): Part 2a: Dose Escalation, D3S-002 and D3S-001 administered orally.
  Part 2b: Dose Expansion, D3S-002 and D3S-001 administered orally.
  Interventions: Drug: D3S-002; Drug: D3S-001

INTERVENTIONS:
Drug: D3S-002 — Oral Tablet
Drug: D3S-001 — Oral Capsule
  Arms: D3S-002 and D3S-001 Combination Therapy

SUMMARY:
This first-in-human (FIH) study aims to assess the safety, tolerability, pharmacokinetics, and recommended phase 2 dose (RP2D) of D3S-002 given orally daily for 21-day cycles in adult subjects with advanced solid tumors with mitogen-activated protein kinase (MAPK) pathway mutations.

ELIGIBILITY:
Inclusion Criteria:

* Part 1: Subjects must have a histologically or cytologically confirmed metastatic or locally advanced solid tumor with evidence of progressive disease.
* Part 2: Subjects must have a histologically or cytologically confirmed metastatic or locally advanced non-small cell lung cancer with evidence of PD.

  * Subjects with non-small cell lung cancer (NSCLC) should have no known epidermal growth factor receptor (EGFR) mutations, ALK/ROS1/RET rearrangements, NTRK1/2/3 gene fusions, v-Raf murine sarcoma viral oncogene homolog B (BRAF) V600E mutations, or MET exon 14 skipping mutations.

Note: EGFR mutations include but are not limited to EGFR Exon19 Deletions, Exon21 p.L858R, Exon21 p.L861Q, Exon18 p.G719X, Exon20 p.S768I, Exon20 Insertions, Exon20 p.T790M. If other EGFR mutations are present, the Investigator should have a consultation with the sponsor's Medical Monitor before making the enrollment decision.

* Part1: Subjects must have documented mitogen-activated protein kinase (MAPK) pathway mutation(s) within the last 5 years identified by a local test on tumor tissue or blood (eg, rat sarcoma (RAS), rapidly accelerated fibrosarcoma (RAF), and MAPK kinase (MAPKK) mutations).
* Part 2: Subject must have documented Kirsten rat sarcoma viral oncogene (KRAS) p. glycine 12 to cysteine (p.G12C) mutation identified within the last 5 years by a local test on tumor tissue or blood.

Note:

• All the local tests should clearly distinguish KRAS p.G12C from all other KRAS p.G12x variants. If not specified, subjects should have no known second KRAS mutations (including G12A, G12V, G12R, G13C, G12D, G12S, H95, Y96, Q61, and R68).

* Part 1: Subjects must be refractory to or intolerable with standard treatment, or have no available standard of care (SOC).
* Part 2: Subject must have received at least 1 line of prior standard of care systemic therapy for locally advanced and unresectable or metastatic disease, including KRAS p.G12C inhibitor.

Note:

* Subjects should only have received 1 type of prior KRAS p.G12Ci treatment (including all types of KRAS p.G12C inhibitor which are either under investigation or in market, except D3S-001).
* During the prior KRAS p.G12C treatment, subject has achieved best response of partial or complete response regardless of KRAS p.G12Ci treatment duration, or stable disease for at least 6 months. However, subjects, who have stopped KRAS p.G12Ci therapy earlier than 6 months due to safety/tolerability reasons only, would be allowed. In such a situation, the Investigator should have a consultation with the Sponsor Medical Monitor before making the enrollment decision.

  * Part 2: Subjects must have measurable disease per RECIST v1.1.
  * Part 2: Subjects must agree to provide archival tumor tissue, if available, for genetic analysis. If archival tumor tissue is not available, or of insufficient quantity, an optional fresh biopsy is highly recommended.
  * Part 2: Subjects must agree to provide blood samples for genetic analysis (Table 2 schedule of activities for Part 2).
  * Subject must have Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
  * Subject must have adequate organ and marrow function within the screening period.
  * Subjects must comply with all reproductive and contraceptive requirements outlined in the protocol.

Exclusion Criteria:

* Subject has any prior treatment with other treatments without adequate washout periods as defined in the protocol.
* Part 2: subjects with mixed small-cell lung cancer, or large cell neuroendocrine histology, or sarcomatoid carcinoma.
* Subject has uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, uncontrolled or significant cardiovascular disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirements, substantially increase risk of incurring AEs, or compromise the ability of the subject to give written informed consent.
* Part 1: Uncontrolled or untreated brain metastasis.
* Part 2: Asymptomatic and stable brain metastases subjects will be eligible for enrollment per the following criteria.

  * Treated or untreated brain metastases
  * Neurologically asymptomatic
  * Stable and not requiring steroids more than 10 mg/day of prednisone or equivalent for at least 4 weeks prior to the first dose of study medication.
* Subject has unresolved treatment-related toxicities from previous anticancer therapy of NCI CTCAE Grade ≥2 (with exception of vitiligo or alopecia).
* Subject has active gastrointestinal disease or other that could interfere significantly with the absorption, distribution, metabolism, or excretion of oral therapy.
* Any concurrent chemotherapy, immunotherapy, targeted therapy, cell therapy, biologic or hormonal therapy and any medical devices for cancer treatment.

NOTE: Other protocol inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | First dose until 30 days after the last dose (or specified in the protocol)
Maximum tolerated dose (MTD) based on Dose limiting toxicities (DLTs) | First dose up to 24 months
Recommended Phase 2 dose (RP2D) | First dose up to 24 months

SECONDARY OUTCOMES:
Part 1: D3S-002 maximum observed plasma concentration (Cmax) | First dose up to 24 months
Part 2: D3S-002 and D3S-001 maximum observed plasma concentration (Cmax) | First dose up to 24 months
Part 1: D3S-002 time to maximum plasma concentration (tmax) | First dose up to 24 months
Part 2: D3S-002 and D3S-001 time to maximum plasma concentration (tmax) | First dose up to 24 months
Part 1: D3S-002 half-life (t1/2) | First dose up to 24 months
Part 2: D3S-002 and D3S-001 half-life (t1/2) | First dose up to 24 months
Part 1: D3S-002 area under the concentration-time curve (AUC) | First dose up to 24 months
Part 2: D3S-002 and D3S-001 area under the concentration-time curve (AUC) | First dose up to 24 months
Objective response rate (ORR) as Determined by the Investigator According to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1) | Until disease progression or end of treatment (up to approximately 24 months)
Disease control rate (DCR) as Determined by the Investigator According to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1) | Until disease progression or end of treatment (up to approximately 24 months)
Progression-free survival (PFS) as determined by the investigator according to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1) | Until disease progression or end of treatment (up to approximately 24 months)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (2):
  - D3 Bio Investigative Site, Detroit, Michigan
  - D3 Bio Investigative Site, New York, New York
- Australia (3):
  - D3 Bio Investigative Site, Blacktown, New South Wales
  - D3 Bio Investigative Site, Bedford Park, South Australia
  - D3 Bio Investigative Site, Nedlands, Western Australia
- China (5):
  - D3 Bio Investigative Site, Beijing, Beijing Municipality
  - D3 Bio Investigative Site, Guangzhou, Guangdong
  - D3 Bio Investigative Site, Harbin, Heilong Jiang
  - D3 Bio Investigative Site, Shanghai, Shanghai Municipality
  - D3 Bio Investigative Site, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No